CLINICAL TRIAL: NCT02040272
Title: Mesothelioma and Radical Surgery 2: a Multicentre Randomised Trial Comparing (Extended) Pleurectomy Decortication Versus no (Extended) Pleurectomy Decortication for Patients With Malignant Pleural Mesothelioma (Mars 2).
Brief Title: Mesothelioma and Radical Surgery 2
Acronym: MARS2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: University of Bristol (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARS2
Record Dates: First submitted 2013-12-20; First posted 2014-01-20 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Experimental): (Extended) pleurectomy decortication
  Interventions: Procedure: (Extended) pleurectomy decortication
- no surgery (No Intervention): no surgery

INTERVENTIONS:
Procedure: (Extended) pleurectomy decortication
  Arms: Surgery

SUMMARY:
Mesothelioma is a cancer of the thin membrane that lines the chest and abdomen. Around 2500 people in the UK are diagnosed with mesothelioma each year and the median survival is approximately 8.5 months. Exposure to asbestos is the most common cause although the cancer does not usually become apparent until 40-60 years after exposure. Anti-cancer drugs (chemotherapy) are usually given to help treat mesothelioma and sometimes lung-sparing surgery (pleurectomy decortication) is undertaken. However, it is not known if this surgery, in addition to chemotherapy, can increase survival and improve the quality of life for patients. The aim of the MARS2 study is to compare surgery - (extended) pleurectomy decortication - with no surgery with respect to overall survival, cost-effectiveness and quality of life. Patients will be followed up by phone at regular intervals for 2 years. Patients will be asked to complete and return a Quality of Life Questionnaire at these time points.

MARS 2 also includes an optional 'Information study', where consenting patients may be interviewed or have their consultations audio-recorded. The aim of the Information study is to explore how a patient makes a decision to take part in research or not, with the overall aim of improving recruitment to clinical trials.

ELIGIBILITY:
Inclusion criteria:

1. 16 years of age or over
2. Tissue (cytology or histology) confirmed epithelioid, sarcomatoid or biphasic mesothelioma
3. Disease confined to one hemi-thorax based on CT assessment
4. Disease deemed surgically resectable
5. Fit for surgery
6. Capacity to provide written informed consent to participate in the trial

Exclusion criteria:

1. Severe shortness of breath (this is defined as an Eastern Cooperative Oncology Group (ECOG) status ≥ 2, or if lung function tests are performed: pre-operative forced expiratory volume after one second (FEV1) or transfer factor of the lung for carbon monoxide (TLco) less than 20%)
2. Serious concomitant disorder that would compromise participant safety during surgery (e.g. evidence of end organ failure)
3. Severe heart failure (this is defined as NYHA III or IV or if an echocardiogram is performed an ejection fraction less than 30%)
4. End stage kidney failure requiring dialysis
5. Liver failure (e.g. encephalopathy and/or coagulation abnormalities)
6. Prisoner
7. Patient lacks capacity to consent
8. Existing co-enrolment in another interventional clinical trial that aims to improve survival

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Survival | 24 months
  The time from randomisation to death will be measured and date of death will be collected on purposely designed case report forms.

SECONDARY OUTCOMES:
Progression free survival to two years | 24 months
Serious adverse health events to two years after randomisation | 24 months
Health Related Quality of Life: EORTC QLQ-C30 (questionnaire) to two years | 24 months
  * 3 types of scales. Functioning scales which include physical functioning, role functioning, emotional function, cognitive functioning and social functioning. Symptom scales which include fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties. An overall global health status/QoL
  * All scales range between 0 and 100.
  * For functioning scales, a high score indicates a high level of functioning. Similarly, a high global health status/QoL score indicates a high quality of life. For symptom scales, a high score indicates a high level of symptoms.
Resource and health service use to two years and during initial surgical admission for surgical arm | 24 months and during initial surgical admission for surgical arm
Health Related Quality of Life: EQ-5D-5L (questionnaire) to two years | 24 Months
  * subscales: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. These range from 1-5.
  * subscales mobility, self-care, usual activities, pain/discomfort, anxiety/depression are combined to calculate an overall index score which ranges from -0.59 to 1.
  * A higher score indicates better quality of life
Health Related Quality of Life: EQ-5D-5L (questionnaire) to two years | 24 months
  * VAS (visual analogue scale) score. Ranges from 0 to 100.
  * A higher score indicates better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lim, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (25):
- United Kingdom (25):
  - Barts Health NHS Trust, London, Whitechapel
  - The Queen Elizabeth Hospital Birmingham, Birmingham
  - North Bristol Trust, Bristol
  - Papworth, Cambridge
  - Colchester, Colchester
  - Derby, Derby
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Golden Jubilee National Hospital, Glasgow
  - Leeds, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Marsden, London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - Wythenshawe, Manchester
  - Clatterbridge, Metropolitan Borough of Wirral
  - South Tees, Middlesbrough
  - South Tyneside NHS Foundation Trust, Newcastle upon Tyne
  - Royal Gwent, Newport
  - Norfolk and Norwich University Hospital, Norwich
  - Oxford University Hospitals, Oxford
  - North West Anglia NHS Foundation Trust, Peterborough
  - University Hospitals Plymouth, Plymouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - New Cross, Wolverhampton

REFERENCES:
- [Derived] Mills N, Farrar N, Warnes B, Ashton KE, Harris R, Rogers CA, Lim E, Elliott D. Strategies to address recruitment to a randomised trial of surgical and non-surgical treatment for cancer: results from a complex recruitment intervention within the Mesothelioma and Radical Surgery 2 (MARS 2) study. BMJ Open. 2024 May 16;14(5):e079108. doi: 10.1136/bmjopen-2023-079108. PMID 38760029
- [Derived] Lim E, Waller D, Lau K, Steele J, Pope A, Ali C, Bilancia R, Keni M, Popat S, O'Brien M, Tokaca N, Maskell N, Stadon L, Fennell D, Nelson L, Edwards J, Tenconi S, Socci L, Rintoul RC, Wood K, Stone A, Muthukumar D, Ingle C, Taylor P, Cove-Smith L, Califano R, Summers Y, Tasigiannopoulos Z, Bille A, Shah R, Fuller E, Macnair A, Shamash J, Mansy T, Milton R, Koh P, Ionescu AA, Treece S, Roy A, Middleton G, Kirk A, Harris RA, Ashton K, Warnes B, Bridgeman E, Joyce K, Mills N, Elliott D, Farrar N, Stokes E, Hughes V, Nicholson AG, Rogers CA; MARS 2 Investigators. Extended pleurectomy decortication and chemotherapy versus chemotherapy alone for pleural mesothelioma (MARS 2): a phase 3 randomised controlled trial. Lancet Respir Med. 2024 Jun;12(6):457-466. doi: 10.1016/S2213-2600(24)00119-X. Epub 2024 May 10. PMID 38740044
- [Derived] Lim E, Darlison L, Edwards J, Elliott D, Fennell DA, Popat S, Rintoul RC, Waller D, Ali C, Bille A, Fuller L, Ionescu A, Keni M, Kirk A, Koh P, Lau K, Mansy T, Maskell NA, Milton R, Muthukumar D, Pope T, Roy A, Shah R, Shamash J, Tasigiannopoulos Z, Taylor P, Treece S, Ashton K, Harris R, Joyce K, Warnes B, Mills N, Stokes EA, Rogers C; MARS 2 Trialists. Mesothelioma and Radical Surgery 2 (MARS 2): protocol for a multicentre randomised trial comparing (extended) pleurectomy decortication versus no (extended) pleurectomy decortication for patients with malignant pleural mesothelioma. BMJ Open. 2020 Sep 1;10(9):e038892. doi: 10.1136/bmjopen-2020-038892. PMID 32873681
- [Derived] Warnock C, Lord K, Taylor B, Tod A. Patient experiences of participation in a radical thoracic surgical trial: findings from the Mesothelioma and Radical Surgery Trial 2 (MARS 2). Trials. 2019 Oct 18;20(1):598. doi: 10.1186/s13063-019-3692-x. PMID 31627746